CLINICAL TRIAL: NCT00143832
Title: Genetic Risk for Attention Deficit Hyperactivity Disorder Expressed in Brain Functioning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Other Study IDs: P03.0465C; METC 04/124
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: fMRI
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Poor inhibitory control has been proposed to be central to the cognitive deficits and symptomatology associated with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a highly heritable disorder with an increased incidence among the siblings of affected individuals. In the current proposal we investigate the expression of genetic susceptibility for ADHD in brain functioning. We will study cognitive functioning in patients with ADHD, their unaffected siblings and healthy matched controls. Our aims are 1) to determine whether increased familial risk for ADHD is associated with differential patterns of brain activation compared to normally developing children, during the performance of tasks designed to probe cognitive functions that are compromised in ADHD and 2) to determine whether differential patterns of activation are similar for boys with ADHD and their unaffected siblings.

DETAILED DESCRIPTION:
Poor inhibitory control has been proposed to be central to the cognitive deficits and symptomatology associated with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a highly heritable disorder with an increased incidence among the siblings of affected individuals. Although studies investigating candidate genes are underway, as yet it remains unclear via which mechanisms the presence of risk genes leads to symptomatology. There is evidence to suggest that individuals at increased genetic risk display some of the cognitive deficits associated with the disorder. In particular poor inhibitory control has been put forward as a potential marker for familial ADHD. Neuroimaging techniques now make it possible to investigate the neural substrate of cognitive deficits associated with psychiatric disorders. Magnetic resonance imaging (MRI) has been used to demonstrate that the neural substrate of cognitive brain function is affected in ADHD. Using a task that taxes inhibitory systems at varying levels of task demands, we demonstrated that increased susceptibility to interference in children with ADHD is paralleled by differences in brain activation, with these children displaying a relative lack of fronto-striatal activation. In a recent study, we demonstrated that the unaffected siblings of patients with ADHD show cortical volumetric deficits, similar to patients themselves. This suggests that individuals at increased risk for ADHD share some of the neural basis of cognitive deficits associated with this disorder. In the current proposal we set out to investigate the expression of genetic susceptibility for ADHD in brain functioning. We will study cognitive functioning in patients with ADHD, their unaffected siblings and healthy matched controls focusing on cognitive control. Our aims are 1) to determine whether increased familial risk for ADHD is associated with differential patterns of brain activation compared to normally developing children, during the performance of tasks designed to probe cognitive functions that are compromised in ADHD and 2) to determine whether differential patterns of activation are similar for boys with ADHD and their unaffected siblings. We intend to include 30 boys with ADHD, 30 of their brothers without ADHD, and 30 matched normal controls in 3 studies focusing on cognitive control and similar cognitive functions that are compromised in ADHD. We will include 10 boys in each group for each study. The proposed studies will utilize variations of a parametric go nogo paradigm previously developed. All subjects will be asked to participate in a functional MR scanning session lasting up to an hour. The whole visit will last a maximum of two hours. There are no known risks associated with MR scanning, therefore this procedure is considered completely safe. By participating in a simulation prior to the scan, we will also minimize anxiety for the subjects. Furthermore, the study will immediately be terminated if a subject becomes anxious, or otherwise indicates that he no longer wishes to participate. All subjects will be offered a gift certificate as a token of appreciation for their effort. In addition, they will be reimbursed for travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 - 20 years
* Male

Inclusion Criteria for Patients with ADHD:

* DSM-IV (APA, 1994) diagnosis of ADHD, according to DISC interview
* Scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form(TRF)
* One brother who meets the inclusion criteria for siblings

Inclusion Criteria for Unaffected Siblings:

* No DSM-IV (APA, 1994) diagnosis according to DISC interview
* No scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)

Inclusion Criteria for Controls:

* No DSM-IV (APA, 1994) diagnosis, according to DISC interview
* No scores in the clinical range on the Child Behavior Checklist (CBCL) and Teacher Rating Form (TRF)

Exclusion Criteria:

* IQ < 70
* Illness of the cardiovascular, the endocrine, the pulmonal or the gastrointestinal system
* Presence of metal objects in or around the body (pacemaker, dental braces)
* History of or present neurological disorder
* For individuals over 12 years of age: legal incompetence, defined as the obvious inability to comprehend the information that is presented by the investigator and is outlined in the Information letter and on which the decision to participate in the study is to be based

Ages: 8 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Durston, Ph.D., Principal Investigator — RMI of Neuroscience, UMC Utrecht; Herman van Engeland, M.D. Ph.D., Study Chair — RMI of Neuroscience, UMC Utrecht
Locations (1):
- Dept. of Child and Adolescent Psychiatry, UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] Durston S, Mulder M, Casey BJ, Ziermans T, van Engeland H. Activation in ventral prefrontal cortex is sensitive to genetic vulnerability for attention-deficit hyperactivity disorder. Biol Psychiatry. 2006 Nov 15;60(10):1062-70. doi: 10.1016/j.biopsych.2005.12.020. Epub 2006 May 19. PMID 16712804
- [Derived] Durston S, Fossella JA, Mulder MJ, Casey BJ, Ziermans TB, Vessaz MN, VAN Engeland H. Dopamine transporter genotype conveys familial risk of attention-deficit/hyperactivity disorder through striatal activation. J Am Acad Child Adolesc Psychiatry. 2008 Jan;47(1):61-67. doi: 10.1097/chi.0b013e31815a5f17. PMID 18174826
- See also: Lab homepage with info for subjects (in Dutch) — http://www.niche-lab.nl